CLINICAL TRIAL: NCT06236555
Title: Exploring 8-iso Prostaglandin F2α and Adenosine Deaminase Levels in Periodontal Health and Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eda Cetin Ozdemir (Other)
Responsible Party: Sponsor-Investigator, Eda Cetin Ozdemir, assistant professor, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023/15, 07
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Periodontal Diseases
Keywords: 8-isoprostane, adenosine deaminase, GCF
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kahramanmaraş Sütçü İmam University (Other): Patients who apply to our clinic for routine periodontal treatment will be included in the study.
  Interventions: Diagnostic Test: 8-iso Prostaglandin F2α and Adenosine Deaminase

INTERVENTIONS:
Diagnostic Test: 8-iso Prostaglandin F2α and Adenosine Deaminase — We took gingival crevicular fluid samples from patients who applied to our clinic and evaluated the -iso Prostaglandin F2α and Adenosine Deaminase levels in the samples.

SUMMARY:
This study aims to assess the diagnostic potential of gingival crevicular fluid (GCF) biomarkers, specifically 8-iso Prostaglandin F2α (8-iso-PGF2α) and adenosine deaminase (ADA), in evaluating periodontal health and disease conditions.

DETAILED DESCRIPTION:
Conducted as a single-blind, cross-sectional investigation, this study comprised 26 individuals categorized as periodontally healthy, 27 with gingivitis, and 27 diagnosed with periodontitis. The participant pool included individuals with various periodontal concerns who were referred to the Department of Periodontology Clinic at Kahramanmaraş Sütçü İmam University. The classification of periodontal health, gingivitis, and chronic periodontitis adhered to the 2018 criteria outlined by the European Federation of Periodontology

ELIGIBILITY:
Inclusion Criteria:

* Patients having more than 20 teeth, minimum age 18, maximum age 65

Exclusion Criteria:

* Patients with systemic disease, Active smokers, Pregnant women, individuals with a history of orthodontic treatment, or those who had undergone periodontal treatment, regardless of whether it was surgical or non-surgical (within the last one year),

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Change in 8-iso Prostaglandin F2α and Adenosine Deaminase scores in periodontal disease | 2023
  We expect 8-iso Prostaglandin F2α and Adenosine Deaminase scores to increase in periodontal disease.

CONTACTS AND LOCATIONS:
Overall Officials: Eda Çetin Özdemir, Dr, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaraş Sütçü İmam University, Kahramanmaraş, Oniki Şubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baltacioglu E, Yuva P, Aydin G, Alver A, Kahraman C, Karabulut E, Akalin FA. Lipid peroxidation levels and total oxidant/antioxidant status in serum and saliva from patients with chronic and aggressive periodontitis. Oxidative stress index: a new biomarker for periodontal disease? J Periodontol. 2014 Oct;85(10):1432-41. doi: 10.1902/jop.2014.130654. Epub 2014 Mar 17. PMID 24635543
- [Background] Barros SP, Williams R, Offenbacher S, Morelli T. Gingival crevicular fluid as a source of biomarkers for periodontitis. Periodontol 2000. 2016 Feb;70(1):53-64. doi: 10.1111/prd.12107. PMID 26662482
- [Background] Basegmez C, Yalcin S, Yalcin F, Ersanli S, Mijiritsky E. Evaluation of periimplant crevicular fluid prostaglandin E2 and matrix metalloproteinase-8 levels from health to periimplant disease status: a prospective study. Implant Dent. 2012 Aug;21(4):306-10. doi: 10.1097/ID.0b013e3182588408. PMID 22814555
- [Background] Basu S. F2-isoprostane induced prostaglandin formation in the rabbit. Free Radic Res. 2006 Mar;40(3):273-7. doi: 10.1080/10715760500511492. PMID 16484043
- [Background] Besada P, Mamedova LK, Palaniappan KK, Gao ZG, Joshi BV, Jeong LS, Civan MM, Jacobson KA. NUCLEOSIDE PRODRUGS OF A3 ADENOSINE RECEPTOR AGONISTS AND ANTAGONISTS. Collect Czechoslov Chem Commun. 2006;71(6):912-928. doi: 10.1135/cccc20060912. PMID 34815583
- [Background] Koregol AC, Kalburgi NB, Kanniappa Sadasivan S, Warad S, Kamat Wagh A, Thomas T, Sinha P. 8-Isoprostane in chronic periodontitis and type II diabetes: Exploring the link. J Dent Res Dent Clin Dent Prospects. 2018 Fall;12(4):252-257. doi: 10.15171/joddd.2018.039. Epub 2018 Dec 19. PMID 30774790